CLINICAL TRIAL: NCT00751543
Title: The Character of Perfusion Parameters Derived From MDCT Between Adenocarcinoma and Squamous Cell Carcinoma of Lung in the Treatment Course of Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeun-Chung Chang / Department of Medical Imaging, National Taiwan University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200705059R
Record Dates: First submitted 2008-09-10; First posted 2008-09-12 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Adenocarcinoma; Squamous Cell Carcinoma; Relevant Condition Terms to the Conditions Field
Keywords: To evaluate the longitudinal change of tumor perfusion in the course of radiation therapy in adenocarcinoma and squamous cell carcinoma using perfusion MDCT; Comparison between adenocarcinoma and squamous cell carcinoma will be evaluated according to the derived perfusion parameter obtained from perfusion MDCT
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: CT, radiation therapy — Computed tomography (CT) is the mainstay for evaluating lung cancer. The advance of multi-row detector CT (MDCT) provides volumetric acquisition within a breath hold, and enables detailed evaluation of tissue and organ perfusion with excellent resolution

SUMMARY:
Lung cancer is one of the leading causes of cancer-related death in Taiwan. Recently, there are more treatment methods available which result in increased patient survival. Although adenocarcinoma and squamous cell carcinoma were both categorized as non-small cell lung cancer (NSCLC), the recent advancement of target therapy implied that these two histologies behave differently (Shah NT, et al. 2005; Sandler A, et al. 2006). Radiation therapy is an important method for locally advanced non-resectable non-small cell lung cancer (NSCLC). Computed tomography (CT) is the mainstay for evaluating lung cancer. The advance of multi-row detector CT (MDCT) provides volumetric acquisition within a breath hold, and enables detailed evaluation of tissue and organ perfusion with excellent resolution. Using this new technique with image post processing, excellent spatial resolution and functional perfusion information can be obtained simultaneously. Therefore, the purpose of this study is to explore not only the longitudinal change of lung cancer eligible for radiation therapy (including concurrent, sequential chemoradiotherapy and high-dose radiation therapy) but also comparison of adenocarcinoma and squamous cell lung cancers using perfusion MDCT. Total twenty patients with histopathologically proved adenocarcinoma or squamous cell carcinoma will be enrolled in this study and receive longitudinal study for perfusion MDCT evaluation before, during radiation therapy and in early and late phases after complete radiation therapy. Dynamic perfusion will be used for processing the image data, and quantitative parameters such as tumor blood volume and permeability etc will be derived. From this study, we expect to understand the change of tumor vascularity after radiation therapy and characters of treatment response of adenocarcinoma and squamous cell carcinoma in addition to the change of tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and up
* Males and females

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
This study will provide information of quantitative measurement of lung cancer, in term of tumor permeability (mL/100 mL/min) and blood volume (mL/100 mL), in addition to tumor size. | Dec, 2008

SECONDARY OUTCOMES:
The information may be beneficial to understand the longitudinal change of internal tumor vascular composition following radiation therapy and between tumors of different histopathology (i.e. adenocarcinoma vs. squamous cell carcinoma). | Dec, 2008

CONTACTS AND LOCATIONS:
Overall Officials: Yeun-Chung Chang, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Yeun-Chung Chang, Taipei, Taiwan, Taiwan